CLINICAL TRIAL: NCT02750969
Title: Lidocaine Patch (Lidocaine 5%) as a Treatment for Tinnitus and Its Accompanied Symptoms
Brief Title: Lidoderm Patch (Lidocaine 5%) for Tinnitus Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15-52
Record Dates: First submitted 2016-03-03; First posted 2016-04-26 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Tinnitus
Keywords: tinnitus; lidocain patch
MeSH Terms: conditions — Tinnitus | interventions — Transdermal Patch; Hearing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. lidoderm patches first (Experimental): 29 tinnitus patients treated first with 3 patches of lidoderm for 1 day, for 12 consecutive hours. 60 hours after removal of the patches the patients will have 3 neutral patches (containing no drug) attach to their back for 12 hours.
  after the removal of each kind of patch the patient will fill 4 types of questionnaires that assess his amount of tinnitus we will compare the questionnaires results before and after the application of those patches.
  Interventions: Device: Lidoderm patch (Lidocaine 5% patch); Procedure: blood test- serum lidocain levels; Other: Hearing tests
- 2. tegaderm patches first (Experimental): 29 tinnitus patients treated first with 3 patches of tegaderm (neutral patch containing no drug) for 1 day, for 12 consecutive hours. 60 hours after removal of the patches the patients will have 3 lidoderm patches attach to their back for 12 hours.
  after the removal of each kind of patch the patient will fill 4 types of questionnaires that assess his amount of tinnitus we will compare the questionnaires results before and after the application of those patches.
  Interventions: Other: Tegaderm patch. (neutral patch, containing no drug); Procedure: blood test- serum lidocain levels; Other: Hearing tests

INTERVENTIONS:
Device: Lidoderm patch (Lidocaine 5% patch) — The investigator will attach the patches on the patient's back for 12 consecutive hours.
  tinnitus questionnaires will be fulfilled by the patient before and after the patches usage . blood test for serum lidocaine level will be measured after the usage of this patch
  Other Names: no other names
  Arms: 1. lidoderm patches first
Other: Tegaderm patch. (neutral patch, containing no drug) — The investigator will attach the patches on the patient's back for 12 consecutive hours.
  tinnitus questionnaires will be fulfilled by the patient before and after the patches usage . blood test for serum lidocaine level will be measured after the usage of this patch
  Arms: 2. tegaderm patches first
Procedure: blood test- serum lidocain levels — each participant will undergo blood test. the participant's group that start the trial with the lidoderm patch and later will use the tegaderm patch will have 2 blood tests for werum lidocain level test. the group taht start the trial with the tegaderm patch and later the lidoderm patch will have only one blood test measuring lidocaine serum level.
  the tubes containing the serum will be shipped abroad via an international medical cargo company for lidocaine levels tests.
Other: Hearing tests — each participant that have not done hearing test in the last 1 year previous to the trial will have one in the first day of the trial.

SUMMARY:
The investigators like to learn whether Lidoderm patch (lidocaine 5%) helps tinnitus patients.

so far it is known that lidocaine I.V do helps tinnitus but until now it is not clear if other means of drug delivery (e.g lidocaine patch) help tinnitus.

The investigators are going to compare 1 day of treatment with lidoderm patch cream Versus (VS.) tegaderm patch (containing no drug) in treating tinnitus patients.

DETAILED DESCRIPTION:
The purpose of the study is to investigate whether lidoderm patch (lidocain 5% patch) cream decreases tinnitus by comparing pretrial questionnaires to post trial questionnaires.

first the investigators are going to invite tinnitus patients for the first visit.

the participants will get full explanation about the trial. in the first visit the investigators will confirm that the participants are suitable for the trial -

1. no exclusion criteria are present
2. the participant will perform 2 screening tests-

   * minimental state examination (MMSE) to evaluate patients cognitive ability to participate in this trial. performance under 24 points is an exclusion criteria
   * Beck depression test- to evaluate patient's ability to be influenced by the lidoderm patch. performance above 24 points is an exclusion criteria the participant will sign on an informed consent form and fulfill a demographic and personal details form.

the participant will undergo ear investigation to exclude ear inflammation, perform audiometry and tinnitus characteristic test to prove sensorineural hearing loss and to get details about the tinnitus characteristics. then the participant will fill 4 questionnaires that reflect the tinnitus loudness and show how much the participant does suffer from this conditions.

1. tinnitus handicap inventory.which estimates the degree that tinnitus affects patients life. it contains 25 questions . The minimum score is 0 and the maximum is 100.
2. Pittsburgh sleep quality index - A 9 questions exam that measures the quality of sleep. the range of results goes between 0-24. The higher the score- the worse is the quality of sleep.
3. visual analogue scale (VAS) for tinnitus subjective loudness evaluation (how much the patient evaluates the loudness of the tinnitus)
4. visual analogue scale (VAS) for tinnitus severity evaluation. (patient's estimation of the amount that tinnitus causes him subjective suffering) Then the investigators will perform randomization: one group will get first the lidoderm patch and later that week the tegaderm patch, the other group will get first the tegaderm patch and later on the lidoderm patch.

Later that day (in the evening), the participant will come to the department (second visit) and the ear nose and throat (ENT) doctor will attach 3 patches on his back for 12 hours (either lidoderm or tegaderm patches).

The participant will be instructed to call the chief investigator When any kind of side effect occurs (topical/ systemic).

in the next morning the participant will come back to our department. (third visit) he will-

1. fill the 4 questionnaires (tinnitus handicap inventory, pittsburgh sleeping scale, VAS severity scale and VAS loudness scale)
2. blood test for lidocaine serum level check will be carried out by a nurse that is authorized to perform blood tests.
3. removal of the patches from the patient's back. 60 hours after the third visit, the participant will attend our department (forth visit). An ENT doctor will attach 3 patches to his back (the second type of patches: participant that had already in the previous visit lidoderm patches will now have the tegaderm patches and vice versa). 12 hours later the participant comes back for his fifth visit. The same 3 steps that were performed in the third visit will be performed again (4 questionnaires, patches removal, blood test for lidocain serum determination).

The investigators hypotheses that lidoderm patches decreases tinnitus as can be estimated by the score of the 4 questionnaires that measure tinnitus aspects.

ELIGIBILITY:
Inclusion Criteria:

* mature (above 18 years old) patients that suffer at least 1 year of tinnitus (unilateral/bilateral

Exclusion Criteria:

* Intermittent/ fluctuative type of tinnitus
* patients that are treated for tinnitus( psychological treatment, hearing aid, drugs, sound generator) or were treated in the last month
* sensitivity to amide anaesthetic
* known hepatic failure
* usage of antiarrhythmic drugs of type 1
* history of seizures
* pregnancy/ lactating
* dermatologic problems in the back
* any patients that develops during the trial local/ systemic symptoms such as rash, pain, itching, fever, nervousness,palpitations will be omitted from the study
* beck depression score of >21
* MMSE test <24

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
questionnaire results change- tinnitus handicap inventory | 1 week: the time between the questionnaire results at the beginning andcompared to the results after using the tegaderm patch and the results after using the lidoderm patch
  tinnitus handicap inventory: estimates the degree that tinnitus affects patients life. It contains 25 questions. The minimum score is 0 and the maximum is 100. The investigators hypotheses that lidoderm patch treatment decreases the score of this questionnaire which means that lidoderm patch improves patients quality of life
questionnaire results- Pittsburgh sleep quality index | 1 week: the time between the questionnaire results at the beginning andcompared to the results after using the tegaderm patch and the results after using the lidoderm patch
  Pittsburgh sleep quality index : A 9 questions exam that measure the quality of sleep. The range of results goes between 0-24. The higher the score - the worse is the quality of sleep. The investigators hypotheses states that lidoderm treatment improves the results of Pittsburgh sleep quality index
tinnitus loudness- visual analogue scale (VAS) | 1 week: the time between the questionnaire results at the beginning andcompared to the results after using the tegaderm patch and the results after using the lidoderm patch
  Tinnitus loudness scale: A range of 1-10 scale. the patient choose which number reflects the loudness of the subjective tinnitus which the patients suffer from. the higher the number- the louder the tinnitus
tinnitus suffer - visual analogue scale (VAS) | 1 week: the time between the questionnaire results at the beginning andcompared to the results after using the tegaderm patch and the results after using the lidoderm patch
  Tinnitus suffer scale: A range of 1-10 scale. the patient choose which number reflects the best the degree in which the tinnitus causes the patient to suffer. the higher the score- the worse is the tinnitus

CONTACTS AND LOCATIONS:
Overall Officials: Avi Shupak, MD, Study Director — "LIN" MEDICAL CENTER
Locations (1):
- Haemek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No